CLINICAL TRIAL: NCT07321678
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of ASC30 Tablets in Participants With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of ASC30 Tablets in Participants With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ascletis Pharma (China) Co., Limited (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC30-203
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ASC30 tablets Dose 1 (Experimental): Participants will receive ASC30 tablets Dose 1 administered orally once daily.
  Interventions: Drug: ASC30 tablets
- ASC30 tablets Dose 2 (Experimental): Participants will receive ASC30 tablets Dose 2 administered orally once daily.
  Interventions: Drug: ASC30 tablets
- ASC30 tablets Dose 3 (Experimental): Participants will receive ASC30 tablets Dose 3 administered orally once daily.
  Interventions: Drug: ASC30 tablets
- Placebo (Placebo Comparator): Participants will receive Placebo administered orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC30 tablets — ASC30 tablets administered orally once daily
  Arms: ASC30 tablets Dose 1; ASC30 tablets Dose 2; ASC30 tablets Dose 3
Drug: Placebo — Placebo administered orally once daily
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled Phase II study is designed to evaluate the efficacy, safety, and tolerability of ASC30 oral tablets formulation in participants with Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes (T2D)
* Have HbA1c ≥7.0% to ≤10.5% as determined by the central laboratory at screening.
* Stable body weight (less than 5% self-reported change within the previous 3 months).
* Have a BMI ≥23.0 kilogram/square meter (kg/m²) at screening.

Exclusion Criteria:

* Have any prior diagnosis of type 1 diabetes mellitus (T1DM), or rare forms of diabetes mellitus
* Have had more than 1 episode of severe hypoglycemia
* Have poorly controlled hypertension
* Have acute or chronic hepatitis and pancreatitis
* Have evidence of a significant active and uncontrolled medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in HbA1c up to 13 weeks in the treatment group compared with the placebo group | Baseline and end of Week 13

SECONDARY OUTCOMES:
Mean change from baseline in fasting blood glucose up to 13 weeks in the treatment group compared with the placebo group | Baseline and end of Week 13
Mean change from baseline in body weight up to 13 weeks in the treatment group compared with placebo group | Baseline and end of Week 13

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Ascletis Clinical Site, Riverside, California
  - Ascletis Clinical Site, San Jose, California
  - Ascletis Clinical Site, Denver, Colorado
  - Ascletis Clinical Site, Miami, Florida
  - Ascletis Clinical Site, Decatur, Georgia
  - Ascletis Clinical Site, Springfield, Missouri
  - Ascletis Clinical Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No